CLINICAL TRIAL: NCT05835466
Title: Phase II Study of Reparixin in Patients With Myelofibrosis Myeloproliferative Neoplasms Research Consortium [MPN-RC 120]
Brief Title: Reparixin in Patients With Myelofibrosis Myeloproliferative Neoplasms Research Consortium (MPN-RC 120)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: Dompé Farmaceutici S.p.A (Industry)
Responsible Party: Principal Investigator, Marina Kremyanskaya, Associate Professor, Icahn School of Medicine at Mount Sinai
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY-22-01764
Record Dates: First submitted 2023-03-29; First posted 2023-04-28 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Myelofibrosis (PMF); Post Essential Thrombocythemia Myelofibrosis (ET-MF); Post Polycythemia Vera Related Myelofibrosis (PV-MF)
MeSH Terms: conditions — Primary Myelofibrosis | interventions — reparixin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Reparixin (Experimental): Eligible patients will receive oral reparixin three times daily on a 4-week cycle for a core study period of 6 cycles (24 weeks). After cycle 6, patients may continue receiving reparixin once daily on a 4-week cycle if at least stable disease (SD) is met by IWG-MRT criteria until loss of response, disease progression, unacceptable toxicity, patient/physician withdrawal, or termination of study by sponsor.
  Interventions: Drug: reparixin

INTERVENTIONS:
Drug: reparixin — reparixin at 1200mg TID three times per day.

SUMMARY:
This is an open label, phase II study to assess the efficacy, safety, and tolerability of Reparixin in patients with DIPSS intermediate-2, or high-risk primary myelofibrosis (PMF), post essential thrombocythemia/polycythemia vera related MF (Post ET/PV MF) after prior treatment, and those who are ineligible or refuse treatment, with a Janus kinase inhibitor (JAKi). 26 patients will be enrolled. Eligible patients will receive oral reparixin three times daily on a 4-week cycle for a core study period of 6 cycles (24 weeks). After cycle 6, patients may continue receiving reparixin once daily on a 4-week cycle if at least stable disease (SD) is met by IWG-MRT criteria until loss of response, disease progression, unacceptable toxicity, patient/physician withdrawal, or termination of study by sponsor.

ELIGIBILITY:
Inclusion Criteria:

* Be ≥ 18 years of age at time of signing the informed consent form (ICF)
* Willing to voluntarily sign the ICF
* Have a pathologically confirmed diagnosis of PMF, post-ET-MF, or post-PV-MF as per the World Health Organization (WHO) diagnostic criteria with intermediate-2 or higher risk disease by DIPSS
* Have an Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2
* Willing to undergo a bone marrow biopsy at screening

  o A bone marrow biopsy obtained within 90 days of screening without intervening treatments and approved by the study chair may suffice.
* Be refractory/resistant to or intolerant of/inappropriate for JAKi therapy as defined by at least one of the following:

  * Treatment for ≥ 3 months with inadequate efficacy as demonstrated by persistent palpable splenomegaly ≥ 5cm or symptoms related to splenomegaly,
  * Treatment for ≥ 28 days complicated by either:
  * Development of a red blood cell transfusion requirement (at least 2 units/month for 2 months)
  * CTCAE grade ≥ 3 AEs of thrombocytopenia, anemia, hematoma, or hemorrhage while being treated with a JAKi
  * Development of non-hematological toxicity that makes patient intolerant of JAKi therapy
  * In the Investigator's judgment, are not candidates for available approved JAKi
* Recovery to ≤ Grade 1 or baseline of any toxicities due to prior systemic treatments, excluding alopecia
* At least two weeks must have elapsed between the last dose of any MF-directed drug treatments or other investigational therapies and start of reparixin

  o Participants may continue hydroxyurea until the day prior to C1D1 if needed for disease control
* Have adequate organ function as demonstrated by the following:

  * ALT (SGPT) and/or AST (SGOT) ≤ 3x upper limit of normal (ULN), or ≤ 4 x ULN (if upon judgment of the treating physician, it is believed to be due to MF-related EMH);
  * Direct bilirubin ≤ 1.5 x ULN; or ≤ 2x ULN (if upon judgment of the treating physician, it is believed to be due to MF-related EMH or documented Gilbert's syndrome);
  * Creatinine clearance ≥ 40 mL/min;
  * Platelet count ≥ 25 x 109/L;
  * Bone marrow and peripheral blood blast count < 10%;
  * ANC ≥ 1000 mm3.
* Life expectancy of at least six months
* Women of childbearing potential (WCBP) and men must agree to use adequate contraception prior to study entry, for the duration of study participation, and for 120 days following completion of therapy. WCBP must also have a negative serum pregnancy test at screening and Cycle 1 Day 1. Should a woman become pregnant or suspect she is pregnant while participating, she should inform her treating physician immediately. (Section 5.9.2)

  o Men must agree to use a condom and not father a child or donate sperm for the duration of the study and for 120 days after the last dose of study therapy
* Ability to adhere to the study visit schedule and all protocol requirements

Exclusion Criteria:

* History of stroke, unstable angina, myocardial infarction, or ventricular arrhythmia requiring medication or mechanical control within the last 6 months
* Other invasive malignancies within the last 3 years, except non-melanoma skin cancer and localized cured prostate and cervical cancer
* Moderate or severe cardiovascular disease meeting one or both of the below criteria:

  * Presence of cardiac disease, including a myocardial infarction within 6 months prior to study entry, unstable angina pectoris, New York Heart Association Class III/IV congestive heart failure, or uncontrolled hypertension
  * Documented major electrocardiogram (ECG) abnormalities (not responding to medical treatments)
* Presence of active serious infection
* Any serious, unstable medical or psychiatric condition that would prevent (as judged by the Investigator) the participant from signing the ICF or any condition, including the presence of laboratory abnormalities, which places the participant at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study
* Participants who have undergone a hematopoietic cell transplant (HCT) within 100 days of the first dose of study therapy, participants on immunosuppressive therapy post-HCT at screening, use of calcineurin inhibitors within 4 weeks prior to first dose of study therapy, or participants with clinically significant graft-versus-host disease (GVHD)

  o Note: The use of topical steroids or < 10mg oral prednisone for ongoing skin GVHD is permitted
* Known history of human immunodeficiency virus (HIV), or known active hepatitis A, B, or C infection
* Impairment of gastrointestinal (GI) function or GI disease that could significantly alter the absorption of reparixin, including any unresolved nausea, vomiting, or diarrhea > CTCAE grade 1
* Is or has an immediate family member (e.g., spouse, parent/legal guardian, sibling, or child) who is investigational site or sponsor staff directly involved with this trial, unless prospective institutional review board (IRB) approval (by chair or designee) is given allowing exception to this criterion for a specific participant
* Organ transplant recipients other than bone marrow transplant
* Women who are pregnant or lactating
* History of splenectomy
* Known hypersensitivity to sulfonamides

  o Hypersensitivity to sulphanilamide antibiotics alone (e.g. sulfamethoxazole) does not qualify for exclusion
* Known hypersensitivity to non-steroidal anti-inflammatory drugs (NSAID), including ibuprofen

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2023-07-24 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Efficacy of reparixin treatment per IWG/ELN criteria | Cycle 6 (each cycle is 4 weeks) Response Assessment
  To estimate the efficacy of reparixin treatment in DIPSS intermediate-2 or high-risk subjects with PMF, post PV-MF, or post ET-MF as assessed by IWG/ELN criteria. The IWG/ELN criteria: CR (complete remission), PR (partial remission), Clinical improvement, Anemia response, Spleen response, Symptoms response, PD (progressive disease), SD (stable disease), Relapse, Cytogenetic remission, and Molecular remission

SECONDARY OUTCOMES:
Response Assessment of IWG/ELN | end of Cycle 6 (each cycle is 4 weeks)
  Response by IWG/ELN criteria at the end of Cycle 6. The IWG/ELN criteria: CR (complete remission), PR (partial remission), Clinical improvement, Anemia response, Spleen response, Symptoms response, PD (progressive disease), SD (stable disease), Relapse, Cytogenetic remission, and Molecular remission
Response Assessment of IWG/ELN | end of Cycle 12 (each cycle is 4 weeks)
  Response by IWG/ELN criteria at the end of Cycle 12. The IWG/ELN criteria: CR (complete remission), PR (partial remission), Clinical improvement, Anemia response, Spleen response, Symptoms response, PD (progressive disease), SD (stable disease), Relapse, Cytogenetic remission, and Molecular remission
Bone marrow fibrosis grade | end of Cycle 6 (each cycle is 4 weeks)
  Bone marrow fibrosis grade at the end of Cycle 6. Bone marrow fibrosis (MF) is graded as MF-0 to MF-3, with higher number indicating more disease.
Bone marrow fibrosis grade | end of Cycle 12 (each cycle is 4 weeks)
  Bone marrow fibrosis grade at the end of Cycle 12. Bone marrow fibrosis (MF) is graded as MF-0 to MF-3, with higher number indicating more disease.
Number of Adverse Events | End of study (24 weeks) plus 3 months
  To assess the safety of reparixin as measured by the adverse event profile of CTCAE v5.0.
Change in Spleen Volume | Baseline and cycle 6 (each cycle is 4 weeks)
  Change in spleen volume by imaging after cycle 6 as compared to baseline spleen volume.
Change in Spleen Volume | Baseline and cycle 12 (each cycle is 4 weeks)
  Change in spleen volume by imaging after cycle 12 as compared to baseline spleen volume.

CONTACTS AND LOCATIONS:
Overall Officials: Marina Kremyanskaya, PhD, MD, Study Chair — Icahn School of Medicine at Mount Sinai; Aaron Gerds, MD, MS, Study Chair — Cleveland Clinic Taussig Cancer Institute
Locations (9):
- United States (9):
  - Moffitt Cancer Center, Tampa, Florida
  - Emory University, Atlanta, Georgia
  - Roswell Park Cancer Institute, Buffalo, New York
  - Ruttenberg Treatment Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - NewYork-Presbyterian/Weill Cornell Medical Center, New York, New York
  - Wake Forest Baptist Health Comprehensive Cancer Center, Winston-Salem, North Carolina
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - The Ohio State University, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: No